CLINICAL TRIAL: NCT06022133
Title: Sodium, Nocturnal Blood Pressure and Nocturnal Pauses in Breathing
Acronym: ROSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesper Norgaard Bech (Other)
Responsible Party: Sponsor-Investigator, Jesper Norgaard Bech, M.D., PhD, head of University Clinic in Nephrology and Hypertension, Regeional Hospital Vest Justland and Aarhus university, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BGH-5-2017; 1-10-72-253-17 (Other: The Scientific Ethical Committees for Central Denmark Region)
Record Dates: First submitted 2020-04-23; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Sodium Imbalance; Nocturnal Blood Pressure; Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Intervention Model Description: Not blinded cross over trial. First arm is usual diet for two weeks, second arm is sodium dietary restriction.
Masking Description: Binding not possible as patients needs to carry out dietary sodium restriction themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary sodium restriction (Experimental): DIetary sodium restriction
  Interventions: Behavioral: Dietary sodium restriction
- Usual diet (No Intervention): Usual diet

INTERVENTIONS:
Behavioral: Dietary sodium restriction — Selfemployed dietary sodium restriction
  Arms: Dietary sodium restriction

SUMMARY:
A reduction of dietary sodium intake reduces blood pressure and risk of cardiovascular disease.

DETAILED DESCRIPTION:
A reduction of dietary sodium intake reduces blood pressure and risk of cardiovascular disease. Patients with hypertension resistant of antihypertensive treatment have a high frequency of non-dipping and obstructive sleep apnoea (OSA). The aim of this project is to analyse the effect of dietary sodium restriction on nocturnal blood pressure and nocturnal pauses in breathing in this patients population.

ELIGIBILITY:
Inclusion Criteria:

* 24h blood pressure > 130/80 mmHg under antihypertensive treatment with three agent, one of these being diuretic. Blood pressure measurement completed after observed intake of antihypertensive medication.
* unchanged antihypertensive treatment for three months
* estimated glomerular function >45 mL/min/1.73 m2

Exclusion Criteria:

* Heart failure assessed from NYHA classification (grade 3-4)
* Presence of clinically significant peripheral edema
* In treatment for obstructive sleep apnea
* Chronic obstructive pulmonary disease (FEV1 <50%)
* Antihypertensive therapy that can not be taken once daily
* Pregnancy or breastfeeding
* Β-albumin <34 g / l
* U-albumin creatinine ratio> 1000 mg / g
* INR> 1.2 (if marevan treatment: ALAT> 200)
* Gluten allergy (dietary guidelines are not adjusted to this group)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in nocturnal systolic blood pressure | from day 14 to day 28
  Comparison of blood pressure measured by 24 hour blood pressure measurements at baseline conditions (after two weeks of usual diet) and intervention (after two weeks of dietary sodium restriction)

SECONDARY OUTCOMES:
Changes in day (systolic and diastolic) and 24h blood pressure (systolic and diastolic) | from day 14 to day 28
  Comparison of blood pressure measured by 24h blood pressure measurements at baseline conditions (after two weeks of usual diet) and intervention (after two weeks of dietary sodium restriction)
Changes in number of nocturnal pauses in breathing (apnoea hypopnoea index, AHI) | from day 14 to day 28
  Comparison of apnoea hypopnoea index measured by cardio respiratory monitoring at baseline conditions (after two weeks of usual diet) and intervention (after two weeks of dietary sodium restriction)
Changes in day:night sodium urinary sodium excretion | from day 14 to day 28
  Comparison of baseline conditions (after two weeks of usual diet) and intervention (after two weeks of dietary sodium restriction)
Changes in urinary excretion of aquaporin-2 (U-AQP2) og epithelial sodium channel (u-ENaCɣ) | from day 14 to day 28
  Comparison of baseline conditions (after two weeks of usual diet) and intervention (after two weeks of dietary sodium restriction)
Changes in endothelial function (nitric oxide (NO), erythrocyte sodium sensitivity) | from day 14 to day 28
  Comparison of biomarkers from blood samples drawn at baseline conditions (after two weeks of usual diet) and intervention (after two weeks of dietary sodium restriction)

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Hornstrup, Principal Investigator — M.D., Ph.D.
Locations (2):
- Denmark (2):
  - University clinic in Nephrology and hypertension, Regional Hospital Godstrup, Gødstrup, Herning
  - Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hornstrup BG, Hoffmann-Petersen N, Lauridsen TG, Bech JN. Dietary sodium restriction reduces blood pressure in patients with treatment resistant hypertension. BMC Nephrol. 2023 Sep 19;24(1):274. doi: 10.1186/s12882-023-03333-9. PMID 37726656